CLINICAL TRIAL: NCT02455050
Title: A Study to Compare a New Eye Drop Formulation With Systane® Gel Drops and Genteal® Lubricant Gel Drops for Moderate to Severe Dry Eye Relief
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11193X-002; NCT02343900 (obsolete NCT alias)
Record Dates: First submitted 2015-01-22; First posted 2015-05-27 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- New Eye Drop Formulation then Systane® (Other): 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks followed by 1 to 2 drops of Systane® Gel Drops in each eye as needed at least 2 times daily for 2 weeks.
  Interventions: Drug: Carboxymethylcellulose Sodium Based Eye Drops; Drug: Systane® Gel Drops
- Systane® then New Eye Drop Formulation (Other): 1 to 2 drops of Systane® Gel Drops in each eye as needed at least 2 times daily for 2 weeks followed by 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks.
  Interventions: Drug: Carboxymethylcellulose Sodium Based Eye Drops; Drug: Systane® Gel Drops
- Genteal® then New Eye Drop Formulation (Other): 1 to 2 drops of Genteal® Lubricant Gel Drops in each eye as needed at least 2 times daily for 2 weeks followed 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks.
  Interventions: Drug: Carboxymethylcellulose Sodium Based Eye Drops; Drug: Genteal® Lubricant Gel Drops
- New Eye Drop Formulation then Genteal® (Other): 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks followed by 1 to 2 drops of Genteal® Lubricant Gel Drops in each eye as needed at least 2 times daily for 2 weeks.
  Interventions: Drug: Carboxymethylcellulose Sodium Based Eye Drops; Drug: Genteal® Lubricant Gel Drops

INTERVENTIONS:
Drug: Carboxymethylcellulose Sodium Based Eye Drops — 1 to 2 drops of Carboxymethylcellulose Sodium Based Eye Drops [New Eye Drop Formula] in each eye.
Drug: Systane® Gel Drops — 1 to 2 drops of Systane® Gel Drops in each eye.
  Other Names: 1 to 2 drops of Systane® Gel Drops in each eye daily.
  Arms: New Eye Drop Formulation then Systane®; Systane® then New Eye Drop Formulation
Drug: Genteal® Lubricant Gel Drops — 1 to 2 drops of Genteal® Lubricant Gel Drops in each eye.
  Arms: Genteal® then New Eye Drop Formulation; New Eye Drop Formulation then Genteal®

SUMMARY:
A study to evaluate the tolerability and acceptability of an investigational eye drop formulation in patients with Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

* Current use of an artificial tear product
* Visual Acuity of at least 20/40 (while wearing glasses, if necessary).

Exclusion Criteria:

* Use of contact lenses in the last 3 months, or anticipated use of contact lenses during the study
* Cataract surgery, laser-assisted in situ keratomileusis (LASIK), photorefractive keratectomy within 6 months
* Use of RESTASIS® Cyclosporine Ophthalmic Emulsion or any topical cyclosporine within 3 months
* Diagnosis of glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Azusa, California, United States

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- New Eye Drop Formulation Then Systane®: 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 1 followed by 1 to 2 drops of Systane® in each eye as needed at least 2 times daily for 2 weeks in Period 2.
- Systane® Then New Eye Drop Formulation: 1 to 2 drops of Systane® Gel Drops in each eye as needed at least 2 times daily for 2 weeks in Period 1 followed by 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 2.
- New Eye Drop Formulation Then Genteal®: 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 1 followed by 1 to 2 drops of Genteal® Lubricant Gel Drops in each eye as needed at least 2 times daily for 2 weeks in Period 2.
- Genteal® Then New Eye Drop Formulation: 1 to 2 drops of Genteal® Lubricant Gel Drops in each eye as needed at least 2 times daily for 2 weeks in Period 1 followed 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 2.
Period: Treatment Period 1
Arm/Group | New Eye Drop Formulation Then Systane® | Systane® Then New Eye Drop Formulation | New Eye Drop Formulation Then Genteal® | Genteal® Then New Eye Drop Formulation
Started | 20 | 19 | 20 | 20
Completed | 19 | 18 | 19 | 18
Not Completed | 1 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2
Period: Treatment Period 2
Arm/Group | New Eye Drop Formulation Then Systane® | Systane® Then New Eye Drop Formulation | New Eye Drop Formulation Then Genteal® | Genteal® Then New Eye Drop Formulation
Started | 19 | 18 | 19 | 18
Completed | 18 | 18 | 17 | 17
Not Completed | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Eye Drop Formulation Then Systane® | Systane® Then New Eye Drop Formulation | New Eye Drop Formulation Then Genteal® | Genteal® Then New Eye Drop Formulation | Total
Number analyzed (Participants) | 20 | 19 | 20 | 20 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.20 (13.41) | 41.79 (15.86) | 40.70 (11.65) | 45.05 (17.05) | 42.95 (14.45)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 15 | 13 | 16 | 58
  Male | 6 | 4 | 7 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Tolerability Survey Score Using a 100 Unit Visual Analog Scale (VAS) in Period 1
Description: Tolerability was assessed using an 8-item survey consisting of 4 positive questions: comfort, soothing, moistening/lubricating and vision clarity and 4 negative questions: stickiness, blur, burning/stinging and discomfort. Participants were instructed to think about their experience over the past week and place a vertical line on the line that best captured how they felt the first 30 minutes after the study drops were administered using the scale: 0 far left of the line to 100 far right on the line. The individual positive scores are added together to obtain the total positive tolerability score from 0 (worst) to 400 (best) and the individual negative scores are added together to obtain the total negative tolerability score for a total possible score of 0 (best) to 400 (worst).
Time Frame: After 14 days of treatment in Period 1 (Follow-up 1 Day 14)
Population: Primary Efficacy Population consisted of all enrolled participants who did not have any significant protocol deviations and completed at least 1 follow-up visit. Participants enrolled in Period 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- New Eye Drop Formulation (Systane® Group); New Eye Drop Formulation (Genteal® Group): 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 1.
- Systane®: 1 to 2 drops of Systane® Gel Drops in each eye as needed at least 2 times daily for 2 weeks in Period 1.
- Genteal®: 1 to 2 drops Genteal® Lubricant Gel drops in each eye as needed at least 2 times daily for 2 weeks in Period 1.
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Positive Questions | 255.74 (119.69) | 280.17 (90.60) | 284.89 (86.18) | 255.83 (94.55)
  Negative Questions | 86.11 (87.83) | 134.89 (97.80) | 101.53 (102.00) | 109.22 (86.33)

2. Primary Outcome: Tolerability Survey Score Using a 100 Unit Visual Analog Scale (VAS) in Period 2
Description: as for outcome 1
Time Frame: After 14 days of treatment in Period 2 (Follow-up 2 Day 35)
Population: Participants from the Primary Efficacy Population, all enrolled participants who did not have any significant protocol deviations and completed at least 1 follow-up visit and participated in Period 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Systane®: 1 to 2 drops of Systane® Gel Drops in each eye as needed at least 2 times daily for 2 weeks in Period 2.
- New Eye Drop Formulation (Systane® Group); New Eye Drop Formulation (Genteal® Group): 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 2.
- Genteal®: 1 to 2 drops Genteal® Lubricant Gel drops in each eye as needed at least 2 times daily for 2 weeks in Period 2.
Arm/Group | Systane® | New Eye Drop Formulation (Systane® Group) | Genteal® | New Eye Drop Formulation (Genteal® Group)
Number analyzed (Participants) | 19 | 18 | 19 | 18
score on a scale
  Positive Questions | 231.33 (112.22) | 295.00 (60.52) | 298.82 (109.15) | 272.12 (125.20)
  Negative Questions | 102.00 (76.69) | 120.00 (71.23) | 54.65 (58.46) | 98.53 (85.60)

3. Secondary Outcome: Ocular Surface Disease Index© (OSDI©) Score Using a 5-Point Scale in Period 1
Description: The OSDI Questionnaire consisted of 12 questions: ocular symptoms (sensitive to light, feel gritty, painful or sore), vision-related functions (blurred vision, poor vision, reading, driving at night, working on a computer and watching TV) and environmental triggers (windy conditions, low humidity/dry areas and air-conditioned areas). Participants were asked to base their evaluation on the frequency of their symptoms over the last week, using a 5-point scale: 0=none of the time to 4=all of time. The total score is converted to a 0 to 100 score where 0 is best and 100 is worst.
Time Frame: Baseline and after 14 days of treatment in Period 1 (Follow-up 1 Day 14)
Population: Primary Efficacy Population consisted of all enrolled participants who did not have any significant protocol deviations and completed at least 1 follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- New Eye Drop Formulation (Genteal® Group): 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 1 or 2.
- Genteal®: 1 to 2 drops Genteal® Lubricant Gel drops in each eye as needed at least 2 times daily for 2 weeks in Period 1 or 2.
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Baseline_Period 1 | 34.76 (13.88) | 36.98 (13.72) | 37.39 (15.99) | 34.79 (10.26)
  Follow-up 1_Day 14 | 27.45 (23.49) | 25.89 (21.07) | 22.85 (25.55) | 23.56 (22.51)

4. Secondary Outcome: Ocular Surface Disease Index© (OSDI©) Score Using a 5-Point Scale in Period 2
Description: as for outcome 3
Time Frame: Baseline and after 14 days of treatment in Period 2 (Follow-up 2 Day 35)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 18 | 19 | 18 | 19
score on a scale
  Baseline_Period 2 | 21.98 (21.85) | 20.36 (24.56) | 18.06 (16.77) | 23.08 (22.15)
  Follow-up 2_Day 35 | 25.88 (24.04) | 21.77 (23.94) | 19.65 (15.60) | 20.42 (22.48)

5. Secondary Outcome: Percentage of Participants Selecting Strongly Agree or Agree in the Acceptability Survey Score Using a 5-Point Scale in Period 1
Description: Acceptability Survey is comprised of 8 questions (Q): Q1-effective dry-eye relief, Q2-eyes feel comfortable, Q3-vision did not blur, Q4-vision normal within 10 minutes, Q5-substantial feel/optimally thick, Q6-eyelashes not matted/crusty, Q7- satisfied overall and Q8-switch to this product/if my doctor recommended. The participant answered the questions using the following scale: a=strongly agree, b=agree, c=neither agree nor disagree, d=disagree and e=strongly disagree. The percentage of participants who selected Strongly Agree or Agree is reported.
Time Frame: After 14 days of treatment in Period 1 (Follow-up 1 Day 14)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
percentage of participants
  Q1_Follow-up 1 Day 14 | 60 | 74 | 75 | 75
  Q2_Follow-up 1 Day 14 | 70 | 74 | 70 | 70
  Q3_Follow-up 1 Day 14 | 35 | 27 | 40 | 30
  Q4_Follow-up 1 Day 14 | 70 | 73 | 85 | 80
  Q5_Follow-up 1 Day 14 | 60 | 79 | 70 | 75
  Q6_Follow-up 1 Day 14 | 55 | 47.3 | 65 | 60
  Q7_Follow-up 1 Day 14 | 60 | 58 | 65 | 65
  Q8_Follow-up 1 Day 14 | 40 | 32 | 60 | 60

6. Secondary Outcome: Percentage of Participants Selecting Strongly Agree or Agree in the Acceptability Survey Score Using a 5-Point Scale in Period 2
Description: as for outcome 5
Time Frame: After 14 days of treatment in Period 2 (Follow-up 2 Day 35)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 18 | 19 | 18 | 19
percentage of participants
  Q1_Follow-up 2 Day 35 | 64 | 60 | 70 | 70
  Q2_Follow-up 2 Day 35 | 79 | 60 | 70 | 70
  Q3_Follow-up 2 Day 35 | 11 | 15 | 20 | 30
  Q4_Follow-up 2 Day 35 | 69 | 70 | 60 | 75
  Q5_Follow-up 2 Day 35 | 52 | 75 | 65 | 60
  Q6_Follow-up 2 Day 35 | 58 | 45 | 55 | 70
  Q7_Follow-up 1 Day 35 | 63 | 50 | 65 | 80
  Q8_Follow-up 2 Day 35 | 52 | 40 | 60 | 75

7. Secondary Outcome: Subjective Evaluation of Symptoms of Dryness (SESoD) Score Using a 5-Point Scale in Period 1
Description: SESoD assessed the severity of dryness (defined as discomfort/irritation due to dry feeling in the eye) evaluated by the participant on a 5-point scale: 0=none, 1=trace, 2=mild, 3=moderate and 4=severe (always notice the symptom and interferes with activities).
Time Frame: Baseline and After 14 days of treatment in Period 1 (Follow-up 1 Day 14)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Baseline_Period 1 | 2.50 (0.89) | 2.21 (0.85) | 2.10 (0.64) | 2.40 (0.82)
  Follow-up 1_Day 14 | 2.26 (1.10) | 1.94 (1.06) | 2.00 (0.82) | 2.28 (0.96)

8. Secondary Outcome: Subjective Evaluation of Symptoms of Dryness (SESoD) Score Using a 5-Point Scale in Period 2
Description: as for outcome 7
Time Frame: Baseline and After 14 days of treatment in Period 2 (Follow-up 2 Day 35)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 18 | 19 | 18 | 19
score on a scale
  Baseline_Period 2 | 1.56 (1.15) | 1.50 (1.15) | 1.67 (0.91) | 1.84 (0.90)
  Follow-Up 2_Day 35 | 1.50 (0.92) | 2.11 (0.68) | 2.24 (0.90) | 1.59 (1.33)

9. Secondary Outcome: Percentage of Participants by Response in End of Study Survey: Assessing Comfort, Blur, and Relief of Symptoms (New Eye Drop Formulation Versus Systane®)
Description: End of Study Survey consisted of 4 questions assessing product preference: Q1-overall comfort, Q2-symptom relief, Q3-less blurring and Q4-preference/willingness to purchase the product. The participant answered each questions using the scale: a=first product better, b=second product better or c=equal. The percentage of participants in each response category is reported.
Time Frame: Day 35
Population: Primary Efficacy Population consisted of all enrolled participants who did not have any significant protocol deviations and completed at least 1 follow-up visit. Data is missing for 3 participants.
Measure: Number; unit: percentage of participants
Groups:
- New Eye Drop Formulation and Systane®: 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 1 or 2 and 1 to 2 drops of Systane® in each eye as needed at least 2 times daily for 2 weeks in Period 1 or 2.
Arm/Group | New Eye Drop Formulation and Systane®
Number analyzed (Participants) | 39
percentage of participants
  Comfort_Prefer New Eye Drop Formulation | 31
  Comfort_Prefer Systane® | 33
  Comfort_Prefer Neither | 28
  Symptom Relief_Prefer New Eye Drop Formulation | 26
  Symptom Relief_Prefer Systane® | 36
  Symptom Relief_Prefer Neither | 31
  Less blurring_Prefer New Eye Drop Formulation | 41
  Less blurring_Prefer Systane® | 31
  Less blurring_Prefer Neither | 21
  Purchase_Prefer New Eye Drop Formulation | 33
  Purchase_Prefer Systane® | 31
  Purchase_Prefer Neither | 28

10. Secondary Outcome: Percentage of Participants by Response in End of Study Survey: Assessing Comfort, Blur, and Relief of Symptoms (New Eye Drop Formulation Versus Genteal®)
Description: as for outcome 9
Time Frame: Day 35
Population: Primary Efficacy Population consisted of all enrolled participants who did not have any significant protocol deviations and completed at least 1 follow-up visit. Data is missing for 6 participants.
Measure: Number; unit: percentage of participants
Groups:
- New Eye Drop Formulation and Genteal®: 1 to 2 drops of New Eye Drop Formulation (carboxymethylcellulose sodium based eye drops) in each eye as needed at least 2 times daily for 2 weeks in Period 1 or 2 and 1 to 2 drops of Genteal® in each eye as needed at least 2 times daily for 2 weeks in Period 1 or 2.
Arm/Group | New Eye Drop Formulation and Genteal®
Number analyzed (Participants) | 40
percentage of participants
  Comfort_Prefer New Eye Drop Formulation | 22
  Comfort_Prefer Genteal® | 42
  Comfort_Prefer Neither | 20
  Symptom Relief_Prefer New Eye Drop Formulation | 22
  Symptom Relief_Prefer Genteal® | 45
  Symptom Relief_Prefer Neither | 18
  Less blurring_Prefer New Eye Drop Formulation | 20
  Less blurring_Prefer Genteal® | 45
  Less blurring_Prefer Neither | 20
  Purchase_Prefer New Eye Drop Formulation | 20
  Purchase_Prefer Genteal® | 45
  Purchase_Prefer Neither | 20

11. Secondary Outcome: Distance Visual Acuity in Period 1
Description: Distance visual acuity is measured in each eye at 5 and 30 minutes post drop instillation using an eye chart at 4 meters and is reported as the number of letters read correctly (ranging from 0 to 100 letters).
Time Frame: After 14 days of treatment in Period 1 (Follow-up 1 Day 14), 5 and 30 minutes post drop instillation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
Letters Read Correctly
  Right Eye (OD)_Follow-Up 1 Day 14_5 Min | 46.05 (9.00) | 46.28 (6.13) | 49.00 (5.98) | 47.44 (6.22)
  OD_Follow-Up 1 Day 14_30 Min | 47.32 (8.84) | 50.78 (4.58) | 51.05 (4.49) | 48.94 (6.40)
  Left Eye (OS)_Follow-Up 1 Day 14_5 Min | 45.84 (7.76) | 47.39 (4.09) | 49.79 (5.63) | 47.78 (5.06)
  OS_Follow-Up 1 Day 14_30 Min | 47.53 (8.59) | 48.44 (4.48) | 50.21 (5.68) | 50.94 (4.05)

12. Secondary Outcome: Distance Visual Acuity in Period 2
Description: as for outcome 11
Time Frame: After 14 days of treatment in Period 2 (Follow-up 2 Day 35), 5 and 30 minutes post drop instillation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters Read Correctly
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 18 | 19 | 18 | 19
Letters Read Correctly
  OD_Follow-Up 2 Day 35_5 Min | 48.56 (5.07) | 46.56 (6.51) | 47.35 (5.70) | 48.65 (5.44)
  OD_Follow-Up 2 Day 35_30 Min | 51.00 (5.81) | 51.11 (5.47) | 50.35 (5.58) | 51.94 (3.49)
  OS_Follow-Up 2 Day 35_5 Min | 48.11 (6.11) | 47.11 (6.28) | 46.47 (7.22) | 49.71 (4.87)
  OS_Follow-Up 2 Day 35_30 Min | 51.11 (5.44) | 49.11 (5.68) | 49.35 (6.01) | 51.24 (3.58)

13. Secondary Outcome: Tear Break-Up Time With Fluorescein in Period 1
Description: Fluorescein was applied to the eyes and three consecutive TBUTs are performed in each eye at 5 and 30 minutes post drop instillation. TBUT is defined as the time (seconds) required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film.
Time Frame: After 14 days of treatment in Period 1 (Follow-up 1 Day 14), 5 and 30 minutes post drop instillation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
seconds
  Right Eye (OD)_Follow-Up 1 Day 14_5 Min | 5.17 (1.89) | 5.45 (2.03) | 4.99 (1.86) | 4.27 (1.03)
  OD_Follow-Up 1 Day 14_30 Min | 6.21 (2.26) | 5.24 (1.56) | 4.86 (1.81) | 5.00 (1.70)
  Left Eye (OS)_Follow-Up 1 Day 14_5 Min | 5.20 (1.93) | 5.39 (1.76) | 5.29 (1.91) | 4.36 (1.30)
  OS_Follow-Up 1 Day 14_30 Min | 6.25 (2.59) | 5.44 (1.94) | 4.89 (1.61) | 4.56 (1.45)

14. Secondary Outcome: Tear Break-Up Time With Fluorescein in Period 2
Description: as for outcome 13
Time Frame: After 14 days of treatment in Period 2 (Follow-up 2 Day 35), 5 and 30 minutes post drop instillation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 18 | 19 | 18 | 19
seconds
  OD_Follow-Up 2 Day 35_ 5 Min | 6.31 (2.58) | 6.13 (2.38) | 4.93 (1.97) | 5.63 (3.49)
  OD_Follow-Up 2 Day 35_30 Min | 5.68 (1.30) | 6.34 (3.00) | 4.94 (1.28) | 5.22 (2.18)
  OS_Follow-Up 2 Day 35_5 Min | 5.64 (2.01) | 6.35 (2.54) | 4.88 (1.44) | 4.74 (2.04)
  OS_Follow-Up 2 Day 35_30 Min | 6.06 (1.57) | 6.01 (1.40) | 5.18 (1.69) | 4.65 (1.27)

15. Secondary Outcome: Eye Drop Experience Survey Score: Assessing Vision, Comfort, and Relief of Symptoms in Period 1
Description: Participants completed the 4 question Eye Drop Experience Survey at 5 and 30 minutes post drop instillation: Question (Q) 1-vision clear/without blur, Q2-drops soothing/comfortable, Q3-drops relieve dry eye symptoms and Q4-comfortable/soothing. Q1 to Q3 were answered using a 5-point scale: 1=strongly disagree to 5=strongly agree. Q4 is answered using a Labeled Hedonic scale by placing a mark on a vertical line where the bottom of the line -100=most uncomfortable/irritating imaginable, middle of the line=neutral to top of the line 100=most comfortable/soothing imaginable.
Time Frame: After 14 days of treatment in Period 1 (Follow-up 1 Day 14), 5 and 30 minutes post drop instillation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 20 | 19 | 20 | 20
score on a scale
  Q1 Follow-up 1 Day 14_5 Minutes (Min) | 3.32 (1.29) | 3.39 (1.24) | 3.58 (1.17) | 3.17 (0.92)
  Q2 Follow-up 1 Day 14_5 Min | 3.53 (1.35) | 3.78 (0.94) | 3.68 (1.00) | 3.72 (0.67)
  Q3 Follow-up 1 Day 14_5 Min | 3.74 (1.10) | 3.61 (0.98) | 3.89 (0.88) | 3.83 (0.86)
  Q4 Follow-up 1 Day 14_5 Min | 26.89 (33.95) | 20.44 (39.04) | 21.11 (27.23) | 28.61 (23.20)
  Q1 Follow-up 1 Day 14_30 Min | 3.84 (1.07) | 4.22 (0.65) | 3.79 (0.98) | 4.28 (0.83)
  Q2 Follow-up 1 Day 14_30 Min | 3.89 (1.10) | 4.22 (0.81) | 4.00 (0.88) | 4.17 (0.38)
  Q3 Follow-up 1 Day 14_30 Min | 3.47 (1.58) | 3.39 (1.24) | 2.84 (1.12) | 3.72 (1.07)
  Q4 Follow-up 1 Day 14_30 Min | 30.05 (34.98) | 43.17 (26.18) | 28.42 (26.05) | 48.06 (21.70)

16. Secondary Outcome: Eye Drop Experience Survey Score: Assessing Vision, Comfort, and Relief of Symptoms in Period 2
Description: as for outcome 15
Time Frame: After 14 days of treatment in Period 2 (Follow-up 2 Day 35), 5 and 30 minutes post drop instillation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Eye Drop Formulation (Systane® Group) | Systane® | New Eye Drop Formulation (Genteal® Group) | Genteal®
Number analyzed (Participants) | 18 | 19 | 18 | 19
score on a scale
  Q1 Follow-up 2 Day 35 _5 Min | 3.22 (1.11) | 3.22 (1.06) | 3.82 (0.81) | 3.76 (0.83)
  Q2 Follow-up 2 Day 35_5 Min | 3.67 (0.97) | 3.28 (0.89) | 3.94 (0.43) | 3.82 (0.81)
  Q3 Follow-up 2 Day 35_5 Min | 3.72 (0.89) | 3.50 (0.92) | 3.88 (0.49) | 4.00 (0.61)
  Q4 Follow-up 2 Day 35_5 Min | 26.89 (29.66) | 18.00 (40.11) | 38.47 (19.01) | 40.06 (30.92)
  Q1 Follow-up 2 Day 35_30 Min | 4.11 (0.76) | 3.94 (1.06) | 4.24 (0.56) | 3.88 (1.05)
  Q2 Follow-up 2 Day 35_30 Min | 3.83 (0.62) | 3.94 (0.94) | 4.24 (0.44) | 4.00 (1.06)
  Q3 Follow-up 2 Day 35_30 Min | 3.89 (0.90) | 3.89 (1.08) | 4.29 (0.59) | 4.06 (1.09)
  Q4 Follow-up 2 Day 35_30 Min | 33.11 (26.87) | 26.00 (36.84) | 47.41 (22.89) | 52.94 (38.02)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 35
Arm/Group | New Eye Drop Formulation Then Systane® | Systane® Then New Eye Drop Formulation | New Eye Drop Formulation Then Genteal® | Genteal® Then New Eye Drop Formulation
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.